CLINICAL TRIAL: NCT06885333
Title: Integrating Whole-Brain Tumor Burden Metrics with Inflammatory and Molecular Markers to Predict Postoperative Neurocognitive Decline in Glioma Patients -a Prospective Cohort Study
Brief Title: Whole-Brain Tumor Burden Metrics with Inflammatory and Molecular Markers to Predict Postoperative Neurocognitive Decline in Glioma
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Simin Zhang, doctor of department of radiology, Principal Investigator, Clinical Professor, West China Hospital
Other Study IDs: 2023745
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Glioma; Glioma : Oligodendroglioma or Astrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Although surgical resection improves overall survival in patients with diffuse Low-grade gliomas (DLGG), it can also result in deterioration of neurocognitive function, which are poorly understood and lack effective predictive models. This study aims to develop a model using whole-brain tumor burden metrics, inflammatory and molecular markers for predicting high risk of neurocognitive decline (ND) postoperatively. The study involved 192 patients with left frontal DLGG. MRI data were analyzed to derive whole-brain tumor burden metrics, including tumor radiomics, whole-brain cortical thickness, myelin content, and network characteristics. postoperative inflammatory and molecular markers were collected. Postoperative follow-up neurocognitive function was assessed using the Montreal Cognitive Assessment at 3 months and 1 year. Machine learning models were constructed using Pycaret.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven DLGG based on 2021 WHO criteria
2. Age ≥ 18 years,
3. Karnofsky Performance Status ≥ 70%,
4. Tumor involved unilateral left frontal lobe and did not reach the central sulcus.

Exclusion Criteria:

1. With previous treatment before image acquisition,
2. Presenting cognitive impairment pre-operatively based on The Montreal Cognitive Assessment (MoCA)
3. Survival of less than 3 months post-surgery
4. Lack of compliance with neurocognitive assessments in 3-month and 1-year after surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 192 glioma patients
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
neurocognitive function was assessed using the Montreal Cognitive Assessment | 3 month
  p neurocognitive function was assessed using the Montreal Cognitive Assessment

IPD SHARING:
Plan to Share IPD: Yes